CLINICAL TRIAL: NCT00230113
Title: A Randomized, Masked, Controlled Study of Omega-3 Polyunsaturated Fatty Acid vs Monounsaturated Fatty Acid Diet Supplementation for the Treatment of Nonalcoholic Fatty Liver Disease
Brief Title: Effect of Omega-3 PUFA Supplementation in NAFLD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Kris Kowdley MD, Virginia Mason Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: DK61728-S2
Record Dates: First submitted 2005-09-29; First posted 2005-09-30 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; NASH; Fatty Liver Disease; Omega-3 Fatty Acid; Fish oil
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Safflower Oil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: Omega-3 fatty acid diet supplementation
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: safflower oil

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid diet supplementation — 4 gm fish oil per day
  Arms: 1
Dietary Supplement: safflower oil — 4 gm per day safflower oil
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether dietary supplementation with omega-3 polyunsaturated fatty acids will decrease the amount of fat in liver.

DETAILED DESCRIPTION:
NAFLD is the most common liver disease in the United States and is also a common cause of abnormal liver tests in the United States. NAFLD includes mild as well as a more severe nonalcoholic fatty liver disease involving liver cell inflammation and damage, called Nonalcoholic Steatohepatitis (NASH). NAFLD is usually discovered because of abnormal liver tests or from a liver ultrasound or CT scan in persons with normal liver enzymes. Liver biopsy may show a mix of fat, inflammation and scarring in the liver. Patients with NAFLD do not drink large amounts of alcohol that can cause this type of liver damage. NAFLD is thought to be related to obesity and diabetes. Unfortunately, there is very little information about important features of NAFLD. These include biochemical, genetic and other features that may help to predict disease progression. The few known risk factors include high blood sugar and lipid levels. Patients with NAFLD often have resistance to the normal action of insulin, a hormone which is important for processing sugar and fat. Increased resistance to insulin leads to fat in the liver. Currently, there is no proven treatment for NAFLD. Several studies in animals suggest that diets containing high levels of omega-3 polyunsaturated fatty acids (PUFA) will decrease the amount of liver fat.

It has long been known that omega-3 fatty acids have several health benefits. For example, a diet rich in these fatty acids reduces the amount of certain fats ("triglycerides") in blood, and might improve the action of the important hormone insulin. Omega-3 fatty acids are contained in certain plant oils (such as canola oil and linseed oil) and marine fish (such as salmon). The purpose of this study is to determine the effect of dietary supplementation with ω-3 polyunsaturated vs monounsaturated fatty acids on intrahepatic fat content in patients with non-alcoholic fatty liver disease as determined by magnetic resonance spectroscopy

ELIGIBILITY:
Inclusion Criteria:

* Acceptance into NASH CRN Database Study
* Exclusion from or unwillingness to participate in the NASH CRN PIVENS Study
* Histological diagnosis or imaging study suggesting NAFLD with at least 20% steatosis
* Willingness to maintain study diet for duration of the study
* At least 18 years of age
* No contraindication for MRI scanning (i.e., pacemaker, shunts etc)

Exclusion Criteria:

* Use of lipid lowering drugs (i.e., statins and fibrate drugs)
* Use of insulin or thiazolidinediones
* Use of drugs possibly associated with NAFLD (amiodarone, methotrexate, systemic glucocorticoids, tetracycline, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, or other known hepatotoxins) for more than 2 consecutive weeks in the 2 years prior to screening
* Initiation of anti-diabetic drugs (insulin, biguanides, sulfonylureas, metformin, thiazolidinediones) in the 3 months prior to randomization
* Initiation of anti-NASH drugs (thiazolidinediones, vitamin E, metformin, UDCA, SAM-e, betaine, milk thistle, gemfibrozil, anti-TNF therapies, probiotics) in the 3 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Reduction of intrahepatic fat content as determined by magnetic resonance spectroscopy | 2 month

SECONDARY OUTCOMES:
Change in serum aminotransferase levels Change in lipid profile Change in levels of proinflammatory cytokines | 2 month
Change in insulin resistance determined by HOMA | 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Kris V Kowdley, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States